CLINICAL TRIAL: NCT07247994
Title: Neurological Manifestations in Children Diagnosed With Inflammatory Bowel Disease in Assiut University Child Hospital
Brief Title: Neurological Manifestations in Children Diagnosed With Inflammatory Bowel Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Bishoy Shehata Fahim (Other)
Responsible Party: Sponsor-Investigator, Bishoy Shehata Fahim, Doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: EIMs in Children with IBD
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: IBD (Inflammatory Bowel Disease)
Keywords: Extraintestinal manifestations; Inflammatory bowel disease; Ibd
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
screen for neurologic and psychiatric disorders in children and

adolescents with IBD.

DETAILED DESCRIPTION:
Neurologic symptoms have a great importance in early diagnosis and

treatment preventing major morbidity and later sequelae, especially if they

precede GI symptoms

The prevalence of neurologic manifestations of IBD varies between 0.2% and

36%. Their pathogenesis of neurologic manifestations in IBD consists of 6

mechanisms: 1.malabsorption and nutritional deficiency 2.metabolic agents

3.infections complicating immune suppression 4.side effects of medications or

iatrogenic as a surgical complication 5.thromboembolism 6.immunological

factors

UC patients are similar to or higher than CD patients in the probability of

neurologic symptoms. Neurologic manifestations and complications include:

headache, dizziness, hypotonia, ADHD, tics, sensory complaints, seizures,

neuropsychiatric disorders, peripherial neuropathy, meningitis, vestibular

dysfunction, idiopathic IC hypertension, cerebral vasculitis, demyelinating

disorders and migraine

ELIGIBILITY:
Inclusion Criteria:

* patients with IBD aged from from 1 to18 years old.

Exclusion Criteria:

* patients with IBD and aged above 18 years old or below 1 year old

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with inflammatory bowel disease in Assiut university child hospital
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Screening for Neurological manifestations among children diagnosed with inflammatory bowel disease in Assiut university children hospital | during the period from January 2026 to January 2027.
  Neurologic symptoms have a great importance in early diagnosis and
  treatment preventing major morbidity and later sequelae, especially if they
  precede GI symptoms
  The prevalence of neurologic manifestations of IBD varies between 0.2% and
  36%. Their pathogenesis of neurologic manifestations in IBD consists of 6
  mechanisms: 1.malabsorption and nutritional deficiency 2.metabolic agents
  3.infections complicating immune suppression 4.side effects of medications or
  iatrogenic as a surgical complication 5.thromboembolism 6.immunological
  factors
  UC patients are similar to or higher than CD patients in the probability of
  neurologic symptoms. Neurologic manifestations and complications include:
  headache, dizziness, hypotonia, ADHD, tics, sensory complaints, seizures,
  neuropsychiatric disorders, peripherial neuropathy, meningitis, vestibular
  dysfunction, idiopathic IC hypertension, cerebral vasculitis, demyelinating
  disorders and migraine
screen for neurologic and psychiatric disorders in children and adolescents with IBD. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nagla Hassan Abufaddan, Professor, Study Director — Assiut university child hospital; Randa Kandeel Abdelaleem, Lecturer, Study Director — Assiut university child hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alsakarneh S, Ahmed M, Jaber F, Abuassi M, Mourad FH, Francis FF, Barada K, Tfayli R, Al-Bawardy B, Farraye FA, Hashash JG. Inflammatory bowel disease burden in the Middle East and North Africa Region: a comprehensive analysis of incidence, prevalence, and mortality from 1990-2019. Ann Gastroenterol. 2024 Sep-Oct;37(5):527-535. doi: 10.20524/aog.2024.0909. Epub 2024 Aug 19. PMID 39238799
- [Result] Kliegman, Nathan J. Blum, Robert C. Tasker, Karen M. Wilson, Joseph W. St Geme, Abigail M. Schuh, Cara L. Mack, Matthew A. Deadorf, Nelson textbook of pediatrics edition 22, Elseveir, vol 2, 2024, pp 2309- 2325.
- [Result] Ben-Or O, Zelnik N, Shaoul R, Pacht A, Lerner A. The neurologic profile of children and adolescents with inflammatory bowel disease. J Child Neurol. 2015 Apr;30(5):551-7. doi: 10.1177/0883073814521296. Epub 2014 Apr 2. PMID 24700662
- [Result] Zhao M, Gonczi L, Lakatos PL, Burisch J. The Burden of Inflammatory Bowel Disease in Europe in 2020. J Crohns Colitis. 2021 Sep 25;15(9):1573-1587. doi: 10.1093/ecco-jcc/jjab029. PMID 33582812
- [Result] Mosli M, Alawadhi S, Hasan F, Abou Rached A, Sanai F, Danese S. Incidence, Prevalence, and Clinical Epidemiology of Inflammatory Bowel Disease in the Arab World: A Systematic Review and Meta-Analysis. Inflamm Intest Dis. 2021 Sep 7;6(3):123-131. doi: 10.1159/000518003. eCollection 2021 Sep. PMID 34722642
- [Result] ulia Gorospe, Joseph Windsor, Lindsay Hracs, Stephanie coward, Michael Buie, Joshua Quan, Lea Caplan, Trends in infammatory bowel disease incidence and prevalence across epidemiologic stages: a global systematic review with meta-analysis, the crohns and colitis foundation and AGA institute, 2024.
- [Result] Gordon H, Burisch J, Ellul P, Karmiris K, Katsanos K, Allocca M, Bamias G, Barreiro-de Acosta M, Braithwaite T, Greuter T, Harwood C, Juillerat P, Lobaton T, Muller-Ladner U, Noor N, Pellino G, Savarino E, Schramm C, Soriano A, Michael Stein J, Uzzan M, van Rheenen PF, Vavricka SR, Vecchi M, Zuily S, Kucharzik T. ECCO Guidelines on Extraintestinal Manifestations in Inflammatory Bowel Disease. J Crohns Colitis. 2024 Jan 27;18(1):1-37. doi: 10.1093/ecco-jcc/jjad108. No abstract available. PMID 37351850
- [Result] Rogler G, Singh A, Kavanaugh A, Rubin DT. Extraintestinal Manifestations of Inflammatory Bowel Disease: Current Concepts, Treatment, and Implications for Disease Management. Gastroenterology. 2021 Oct;161(4):1118-1132. doi: 10.1053/j.gastro.2021.07.042. Epub 2021 Aug 3. PMID 34358489